CLINICAL TRIAL: NCT03797261
Title: Phase 1b Study of Venetoclax and AMG 176 in Patients With Relapsed/Refractory Hematologic Malignancies
Brief Title: A Study of Venetoclax and AMG 176 in Patients With Relapsed/Refractory Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-785; 2018-003314-41 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Acute Myeloid Leukemia; Non-Hodgkin's Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: Acute Myeloid Leukemia; Non-Hodgkin's Lymphoma; Cancer; Venetoclax; AMG 176; diffuse large B-cell lymphoma (DLBCL)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Neoplasms | interventions — venetoclax; tapotoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + AMG 176 (Experimental): Venetoclax and AMG 176 will be administered in combination. Different combinations of dose levels for venetoclax and AMG 176 will be explored.
  Interventions: Drug: Venetoclax; Drug: AMG 176

INTERVENTIONS:
Drug: Venetoclax — tablet, oral
  Other Names: ABT-199
Drug: AMG 176 — solution, intravenous

SUMMARY:
This dose-escalation study evaluating the safety, pharmacokinetics and preliminary efficacy of venetoclax in combination with AMG 176 in participants with relapsed or refractory acute myeloid leukemia (AML) and participants with Non-Hodgkin's lymphoma (NHL)/diffuse large B-cell lymphoma (DLBCL).

This study will include a dose escalation phase to identify the maximum tolerated dose/recommended phase 2 dose (MTD/RPTD) of venetoclax plus AMG 176 as well as a dose expansion phase to confirm safety, explore efficacy, and confirm the suitability of the preliminary RPTD.

ELIGIBILITY:
Inclusion Criteria:

* Adequate kidney, liver and hematology values as described in the protocol.
* Diagnosis of relapsed or refractory (R/R) acute myeloid leukemia (AML) or R/R Non-Hodgkin's lymphoma (NHL)/diffuse large B-cell lymphoma (DLBCL) confirmed by the World Health Organization (WHO) criteria, as appropriate.
* Meets the following disease activity criteria:
* AML: must have received at least 1 prior therapy for AML and be ineligible for cytotoxic therapy and allogeneic stem cell transplant.
* NHL/DLBCL: measurable disease with a bidimensional lesion measuring at least 1.5 cm; received at least 1 prior therapy for NHL with no curative treatment option as determined by the investigator and be ineligible for a stem cell transplant.

Exclusion Criteria:

* History of clinically significant medical condition that, in the opinion of the investigator, would adversely affect participation in this study.
* History of of any malignancy within the last 6 months except for those specified in this protocol and low-grade malignancies not requiring active treatment such as non-melanoma skin cancer, cervical intraepithelial neoplasia, or prostate cancer in situ.
* Prior allogeneic stem cell transplant or autologous stem cell transplant within 100 days of study drug administration and no signs or symptoms of acute or chronic graft-versus-host disease.
* Previous enrollment in a randomized trial including either venetoclax or AMG 176.
* Known active or chronic pancreatitis; severe chronic obstructive pulmonary disease with hypoxemia; central nervous system manifestations of malignancy.
* Active, uncontrolled infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RPTD) for Venetoclax + AMG 176 | Up to 28 days after first dose of study drug in a dose-escalation phase
  The MTD and/or RPTD of venetoclax and of AMG 176 will be determined during the dose escalation phase of the study.
Number of Participants With Adverse Events | From first dose of study drug until 30 days or 5 half-lives after discontinuation of study drug administration will be collected (up to approximately 4 years).
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Composite Complete Remission Rate (CRc) for Participants with AML | Up to approximately 2 years from last subject first dose
  CRc rate is defined as CR + CRi (CR with incomplete blood count recovery).
Objective Response Rate (ORR) for Participants with AML | Up to approximately 2 years from last subject first dose
  ORR is defined as the percentage of participants with documented partial response (PR) or better (CR + CRi + partial response [PR]) based on International Working Group (IWG) criteria for AML
ORR for Participants with NHL | Up to approximately 2 years from last subject first dose
  ORR is defined as the percentage of participants with documented CR + PR based on Lugano criteria for NHL.
Maximum Plasma Concentration (Cmax) of Venetoclax | Up to approximately 28 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of venetoclax.
Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax | Up to approximately 28 days after first dose of study drug
  Time to maximum plasma concentration (Tmax) of Venetoclax.
AUC of Venetoclax | Up to approximately 28 days after first dose of study drug
  Area under the plasma concentration-time curve (AUC) of venetoclax.
Maximum Plasma Concentration (Cmax) of AMG 176 | Up to approximately 16 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of AMG 176
Half-life (t1/2) of AMG 176 | Approximately 16 days after first dose of study drug
  Terminal phase elimination half-life (t1/2)
AUC of AMG 176 | Approximately 16 days after first dose of study drug
  Area Under the Plasma Concentration-time Curve (AUC) of AMG 176
Clearance (CL) of AMG 176 | Approximately 16 days after first dose of study drug
  Clearance (CL) is defined the volume of plasma cleared of the drug per unit time.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (17):
- United States (9):
  - City of Hope /ID# 207393, Duarte, California
  - USC Norris Cancer Center /ID# 207396, Los Angeles, California
  - University of Iowa Hospitals and Clinics /ID# 207459, Iowa City, Iowa
  - Univ Kansas Med Ctr /ID# 207480, Kansas City, Kansas
  - Duplicate_Dana-Farber Cancer Institute /ID# 207367, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 206995, St Louis, Missouri
  - NYU Langone Medical Center /ID# 207390, New York, New York
  - Unc /Id# 207388, Chapel Hill, North Carolina
  - UPMC Hillman Cancer Ctr /ID# 208482, Pittsburgh, Pennsylvania
- Australia (3):
  - Calvary Mater Newcastle /ID# 211455, Waratah, New South Wales
  - Royal Adelaide Hospital /ID# 210602, Adelaide, South Australia
  - Alfred Health /ID# 210350, Melbourne, Victoria
- Germany (5):
  - Universitaetsklinikum Frankfurt /ID# 207984, Frankfurt am Main, Hesse
  - Universitaetsklinikum Leipzig /ID# 209824, Leipzig, Saxony
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 207987, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 207803, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 207788, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com